CLINICAL TRIAL: NCT04543474
Title: Treatment Efficacy of a Low FODMAP Diet Compared to a Low Lactose Diet in IBS Patients: a Randomized, Cross-over Designed Study
Brief Title: Treatment Efficacy of Low FODMAP Versus Low Lactose Diet in IBS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Claudia Krieger-Grübel, Principal Investigator, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 130225
Record Dates: First submitted 2020-08-15; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients starting with a low lactose diet for 3 weeks, followed by a wash out phase of 3 week, before crossing over to the low FODMAP diet for 3 weeks
  Interventions: Other: Low Lactose Diet; Other: Low FODMAP Diet
- Group 2 (Active Comparator): Patients starting with a low FODMAP diet for 3 weeks, followed by a wash out phase of 3 week, before crossing over to the low lactose diet for 3 weeks.
  Interventions: Other: Low Lactose Diet; Other: Low FODMAP Diet

INTERVENTIONS:
Other: Low Lactose Diet — First, there was a run-in period (day 1-14), during which patients were randomly assigned by computer-generated bloc randomization to either the LLD or the LFD for 21 days (day 15-35). A dietician educated the participants on the first interventional diet. This phase was followed by a wash-out period of 21 days (day 36-56) with resumption of a normal balanced daily-life diet before crossing over to the alternate interventional diet (day 57-77). There were visits at the end of the washout phase with an instruction on the second interventional diet and at the end of the study.
Other: Low FODMAP Diet — First, there was a run-in period (day 1-14), during which patients were randomly assigned by computer-generated bloc randomization to either the LLD or the LFD for 21 days (day 15-35). A dietician educated the participants on the first interventional diet. This phase was followed by a wash-out period of 21 days (day 36-56) with resumption of a normal balanced daily-life diet before crossing over to the alternate interventional diet (day 57-77). There were visits at the end of the washout phase with an instruction on the second interventional diet and at the end of the study.

SUMMARY:
A low FODMAP diet (LFD) has become a standard treatment in irritable bowel syndrome (IBS) patients. Compliant adherence to a LFD is challenging. The investigator looked at the effect of a LFD compared to a less restrictive low lactose diet (LLD) in a randomized cross-over trial with IBS patients.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic gastrointestinal disorder. It affects 10 - 20% of the adult population. Pharmaceutical therapy as bulking agents, anticholinergics, antispasmodics, and antidiarrheals are mostly unsatisfactory and many gastroenterologists recommend therefore dietary management. Most patients note that various foods elicit abdominal symptoms and therefore restrict their diet .

The low fermentable oligosaccharide, disaccharide, monosaccharide and polyol (FODMAP) diet has currently the greatest evidence for efficacy in IBS. The rationale behind the LFD is the exclusion of poorly absorbed short-chain carbohydrates which would create an osmotic load, drag fluid into the small intestine and would be fermented by the colonic microbiome, both leading to abdominal distention and increased luminal influx. FODMAPs do not cause symptoms in healthy adults as they neither show these abnormalities in gut physiology nor suffer from visceral hypersensitivity .

It is not known however whether change in symptoms is induced by a reduction in all FODMAPs or simply a single component as for example lactose. If there is a lactase deficiency, as it is the case in 2-20% of Central- / Northern Europeans, lactose cannot be hydrolysed and causes the above mentioned symptoms. Many IBS patients avoid lactose, even though only few have a lactase deficiency. Lactose intolerance but not lactase deficiency is more frequent in patients with IBS. The investigator wanted to examine if the demanding LFD is more effective than elimination of lactose alone.

Our study, comparing in detail the effects of low FODMAP versus low lactose diet in IBS patients is a novelty, analysing a clinically highly relevant topic.

ELIGIBILITY:
Inclusion Criteria:

* functional bowel symptoms as defined by the Rome IV criteria
* subjective lactose intolerance

Exclusion Criteria:

* pharmacologic agents to alter symptoms (laxatives, antidiarrheal agents)
* smoking
* antibiotic therapy within the last 4 weeks
* gastrointestinal diseases (Celiac disease was excluded by negative serologic testing while on a gluten containing diet
* any type of food allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Change from gastrointestinal symptoms in Irritable Bowel Syndrome (IBS symptom severity score) from Baseline to "post intervention diet". | The IBS SSS was assessed at the end of the run in period and at the end of the intervention diets (low lactose and low FODMAP diet) at day 14, 35 and 77.
  The symptom severity score (IBS-SSS) is a validated score to evaluate the severity of an IBS. The five subscores for abdominal pain (severity and frequency), abdominal distension, satisfaction with stool habits and interference of IBS with daily life were each rated on a VAS (visual analogue scale) 0-100 mm scale and added up to a maximal sum of 500. A total score of 75 - 175 was regarded as mild, 175 - 300 as moderate and > 300 as severe IBS.

SECONDARY OUTCOMES:
IBS symptom severity subscore "abdominal pain severity" | IBS subscores were assesses at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77.
  The subscore (abdominal pain severity was assessed individually, on a VAS (visual analogue scale) 0-100 mm scale (the less, the better)
IBS- symptom severity subscore "abdominal pain frequency" | IBS subscores were assesses at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77.
  The subscore abdominal pain frequency was assessed individually on a VAS (visual analogue scale) 0-100 mm scale (the less, the better)
IBS- symptom severity subscore "abdominal distension" | IBS subscores were assesses at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77.
  The subscore abdominal distension was assessed individually on a VAS (visual analogue scale) 0-100 mm scale (the less, the better)
IBS symptom severity subscore "satisfaction with stool habits" | IBS subscores were assesses at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77.
  The subscore satisfaction with stool habits was assessed individually on a VAS (visual analogue scale) 0-100 mm scale (the less the better).
IBS symptom severity subscore "interference of IBS with daily life" | IBS subscores were assesses at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77.
  The subscore satisfaction with stool habits was assessed individually on a VAS (visual analogue scale) 0-100 mm scale (the less, the better)
IBS symptom severity score | IBS SSS (total) was assessed at the end of the run-in (day 14), and wash-out phase (day 56).
  The symptom severity score (IBS-SSS) is a validated score to evaluate the severity of an IBS. The five subscores for abdominal pain (severity and frequency), abdominal distension, satisfaction with stool habits and interference of IBS with daily life were each rated on a VAS 0-100 mm scale and added up to a maximal sum of 500. A total score of 75 - 175 was regarded as mild, 175 - 300 as moderate and > 300 as severe IBS.
Stool frequency | Stool frequency was assessed daily throughout the study (day 1-77).
  Patients recorded stool frequency
Stool consistency | Stool consistency was assessed daily throughout the study (day 1-77).
  Patients recorded stool consistency according to the Bristol Stool Chart (BSC) Type 1 hard lumps, Type 2 sausage shaped but lumpy, Type 3 sausage with cracks, Type 4 smooth sausage, Type 5 soft blobs, Type 6 fluffy pieces, Type 7 entirely liquid.
Body weight | Body weight was assesses at the beginning of the study (day 1) and at the end of each trial phase (run-in, first intervention diet, wash-out, second intervention diet) at day 14, 35, 56 and 77).
  Body weight in kg.

IPD SHARING:
Plan to Share IPD: No